CLINICAL TRIAL: NCT06742398
Title: Running Performance in Response to Different Forms of Carbohydrate
Brief Title: Carbohydrates and Running Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Professor and Department Head, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PROJECT00005235
Record Dates: First submitted 2024-12-13; First posted 2024-12-19 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: For the three testing visits (V2-V4), subjects will perform a 12.8 km running TT on a motorized treadmill, with the only difference between visits being the form of treatment. Either a carbohydrate MR solution (called CMR), water MR solution as a control (called WMR), or carbohydrate DS (called DS) will be administered at each visit in a randomized order. Study visits will be separated by at least 5 days, and all visits will take place in the Human Nutrition Lab (HNL) at the University of Georgia in Athens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate Mouth Rinse (Active Comparator): Subjects will be instructed to complete the 12.8 km time trial (TT) as quickly as possible. They will be able to adjust the speed on the treadmill throughout the TT but will have no knowledge of what speed they are actually running at. The researcher will monitor the progress of the TT, and the completion time will be recorded. The carbohydrate mouth rinse treatment will be given just before the start of the TT and every 12.5% of the TT, but not after the completion of the TT.
  Interventions: Other: Carbohydrate Mouth Rinse
- Water Mouth Rinse (Sham Comparator): Subjects will be instructed to complete the 12.8 km time trial (TT) as quickly as possible. They will be able to adjust the speed on the treadmill throughout the TT but will have no knowledge of what speed they are actually running at. The researcher will monitor the progress of the TT, and the completion time will be recorded. The water mouth rinse treatment will be given just before the start of the TT and every 12.5% of the TT, but not after the completion of the TT.
  Interventions: Other: Water Mouth Rinse
- Carbohydrate Dissolvable Strip (Experimental): Subjects will be instructed to complete the 12.8 km time trial (TT) as quickly as possible. They will be able to adjust the speed on the treadmill throughout the TT but will have no knowledge of what speed they are actually running at. The researcher will monitor the progress of the TT, and the completion time will be recorded. The carbohydrate dissolvable strip treatment will be given just before the start of the TT and every 12.5% of the TT, but not after the completion of the TT.
  Interventions: Other: Carbohydrate Dissolvable Strip

INTERVENTIONS:
Other: Carbohydrate Dissolvable Strip — Participants are provided with a carbohydrate dissolvable strip for every 12.5% of the time trial that is completed (calculated based on the distance covered).
  The carbohydrate dissolvable strip (Innsol Health Corp.) is primarily composed of sucrose and glucose; however, the full ingredient list includes pullulan, mannitol, menthol, hydroxyl propyl methyl cellulose, eucalyptol, polysorbate 80, glyceryl oleate, purified water.
  Arms: Carbohydrate Dissolvable Strip
Other: Carbohydrate Mouth Rinse — Participants are provided with a carbohydrate mouth rinse for every 12.5% of the time trial that is completed (calculated based on the distance covered).
  The sucrose solution will consist of 64g of sucrose dissolved in 1000 mL of water, with a bolus of 25 mL being used for each mouth rinse. Each mouth rinse solution will have 2mL of red food dye FD&C Red No. 40 to ensure the same sensory response through appearance.
  Arms: Carbohydrate Mouth Rinse
Other: Water Mouth Rinse — Participants are provided with a water mouth rinse for every 12.5% of the time trial that is completed (calculated based on the distance covered).
  The water solution will consist of 1000 mL of water, with a bolus of 25 mL being used for each mouth rinse. Each mouth rinse solution will have 2mL of red food dye FD&C Red No. 40 to ensure the same sensory response through appearance.
  Arms: Water Mouth Rinse

SUMMARY:
Carbohydrates serve as the body's primary energy source during intense exercise, and consuming carbohydrates during exercise has been shown to improve exercise performance. Previous research has shown that the presence of carbohydrates in the mouth activates sweet taste receptors on the tongue, which signal the brain to increase neural activation in areas associated with motor functioning, sensory perception, and reward centers during exercise through this CPR. The primary objective of this intervention is to establish how carbohydrates delivered in different forms (MR versus dissolvable strip (DS)) affect running performance during a 12.8km running TT.

DETAILED DESCRIPTION:
This trial will be a randomized, controlled crossover design in humans. There will be four study visits (see Figure 1 below). The first visit (Baseline Visit/V1) will entail signing informed consent documents, anthropometric measurements, familiarization with the MR and DS, and the exercise protocol. For the three testing visits (V2-V4), subjects will perform a 12.8 km running TT on a motorized treadmill, with the only difference between visits being the form of treatment. Either a carbohydrate MR solution (called CMR), water MR solution as a control (called WMR), or carbohydrate DS (called CDS) will be administered at each visit in a randomized order. Study visits will be separated by at least 5 days, and all visits will take place in the Human Nutrition Lab (HNL) at the University of Georgia in Athens.

Specific Aims:

1. To examine the effect of carbohydrates delivered in different forms on running performance.
2. To examine the effect of carbohydrates delivered in different forms on physiologic measures as well as perceived exertion.

Hypotheses:

1. The investigators hypothesize that the carbohydrate-containing MR and DS will result in faster TT performance compared to a water MR (control).
2. The Investigators hypothesize that the carbohydrate-containing DS and MR will elicit higher HR and blood lactate levels (indicating greater levels of intensity) compared to control without significantly increasing RPE during the running TT.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Male or Female
* Normal body mass index (BMI) between 18.0-24.9kg/m2
* All subjects will be endurance-trained athletes who participate in training on a regular basis (≥4 sessions per week for at least 1 hour per session of aerobic/endurance exercise (such as running, cycling, or swimming)
* Women will be tested only during the follicular phase of their menstrual cycle (days 2-9) to control for any fluctuation in hormones
* Individuals aged 35 or older must pass the Physical Activity Readiness Questionnaire (PARQ2)

Exclusion Criteria:

* Anyone eating a low carbohydrate diet (such as The Zone™ Diet or Atkins™ Diet)
* Changes in current exercise program
* Chronic diseases (including but not limited to type II diabetes, hypertension, hypotension, hyperthyroidism, cardiovascular disease, and cancer)
* Medications that could alter metabolic rate or hydration status
* Supplement use other than fish oil or vitamin/mineral supplements
* Nicotine use
* Pregnancy or nursing
* Donation of blood in the 20 days prior to testing
* A failing result on the Physical Activity Readiness Questionnaire (PARQ2) for those aged 35 or older
* Allergy to red food dye FD&C Red No. 40

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Completion Times | Baseline/start time to approximately 1.5 hours
  Measured by the time it takes from the beginning of the time trial (0.0 km) to finish the 12.8 km distance (minutes and seconds).
Percent Change in Completion Time from Control | Baseline/start time to approximately 1.5 hours
  Measured by subtracting the completion time of the experimental and active comparator treatments from the control/sham comparator and dividing by the control/sham comparator, then multiplying by 100 to convert to a percentage (percent change in completion time from control).
Mile Pace Splits During the Time Trial | Baseline/start time to approximately 1.5 hours
  Measured by the time it takes to complete each individual 12.5% increment of the total 12.8 km time trial (minutes and seconds).
Blood Lactate Levels | Baseline to approximately 1.5 hours
  The blood lactate concentration immediately before beginning and after completion of the time trial at visits 2-4 (mmol/L).
Ratings of Perceived Exertion | Baseline/start time to approximately 1.5 hours
  The Borg's Rating of Perceived Exertion scale will be used to measure self-reported perceived exertion (RPE) ratings. The sale minimum is 6, and the maximum is 20. Higher scores indicate higher feelings of exertion.
Maximum Heart Rate | Baseline/start time to approximately 1.5 hours
  A continuous heart rate monitor (Polar H9 Heart Rate Sensor) will measure maximum heart rate (beats per minute).
Change in Time Trial Heart Rate Values | Change from baseline/start time to approximately 1.5 hours
  A continuous heart rate monitor (Polar H9 Heart Rate Sensor) will be used to measure heart rate throughout the time trial (beats per minute).
Percent Change in Blood Lactate Pre-to-Post Time Trial | Percent change from baseline/start time to approximately 1.5 hours
  Measured by subtracting post-blood lactate from pre-blood lactate and dividing by pre-blood lactate, then multiplying by 100 to convert to a percentage (percent change in lactate).

SECONDARY OUTCOMES:
Body Weight Pre-to-Post Time Trial | Baseline/start time to approximately 1.5 hours
  Body weight (kg)
Acute Dietary Intake | Day before visit 2, Day before visit 3, Day before visit 4
  One-day food logs will be used to record all foods and beverages consumed the day before testing days.
Subjective Sensory Feelings by Treatment | At the end of each testing visit (days 1-3)
  Subjective feelings related to the sweetness, saltiness, sourness, bitterness, savories, and pleasantness of intervention food are measured by visual analog scales (mm) and generalized labeled magnitude scales (mm). Both scales are measured from 0-100 mm. Higher ratings indicate higher sensory scores.

OTHER OUTCOMES:
Five-Point Just-About-Right Scale | At the end of each testing visit (days 1-3)
  The Five-Point Just-About-Right Scale will be used to measure the appropriateness of each treatment according to consumer perception. The scale is measured from 1 to 5. Higher ratings indicate strong perceptions of the treatment.
Consumer Product Questionnaire | At the end of the final testing visit (day 3 of intervention)
  A Consumer Product Questionnaire will assess various consumer experiences and perceptions regarding the dissolvable strip and Mouth rinse treatments. This questionnaire contains "yes or no" questions regarding nutrition supplementation and asks about consumer experiences if any past supplements have been used.
Net Promotor Score Rating | At the end of the testing visit in which the participants received the dissolvable strip (day 1, 2, or 3)
  A Net Promoter Score Questionnaire will be used to measure satisfaction by asking how likely it is that consumers would recommend the dissolvable strip product to a friend or colleague. The scale used goes from 1 to 10; the higher the score indicates an increased likeliness of recommending the product to a friend or colleague.
New Product Questionnaire Rating | At the end of the testing visit in which the participants received the dissolvable strip (day 1, 2, or 3)
  A New Product Questionnaire will be used to measure various aspects such as market needs, product features, customer preferences, usage patterns, competitor analyses, pricing, purchase intent, and improvement suggestions to gather insights and feedback about the dissolvable strip product. The scale used goes from 1 to 5, and the greater the number, the worse the feeling about the product.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie A Cooper, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No